CLINICAL TRIAL: NCT00087360
Title: Providing Genetic And Environmental Cancer Risk Assessment In Primary Care
Brief Title: Genetic and Environmental Risk Assessment for Colorectal Cancer in Healthy Participants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fox Chase Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Screening
Other Study IDs: FCCC-03030; CDR0000374972 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2004-07-08; First posted 2004-07-12 (Estimated); Last update posted 2013-07-11 (Estimated); Status verified 2013-07

CONDITIONS: Colorectal Cancer
Keywords: colon cancer; rectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — Counseling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: counseling intervention
Other: physiologic testing
Procedure: evaluation of cancer risk factors

SUMMARY:
RATIONALE: Evaluating the knowledge and attitudes of healthy participants toward a new diet and gene test for colorectal cancer risk may help doctors improve acceptance of colorectal cancer screening.

PURPOSE: This clinical trial is studying the knowledge and attitudes of healthy participants toward genetic and environmental risk assessment for colorectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Part 1

* Determine the willingness of healthy participants to enroll in a genetic and environmental risk assessment for colorectal cancer.
* Determine the impact of decision counseling on knowledge and attitudes about genetic and environmental risk assessment (GERA) and colorectal cancer screening in these participants.
* Determine participants' understanding of GERA.
* Determine participants' response to GERA results.

Part 2

* Determine awareness of, and interest in, diet and genetic assessment for colorectal cancer among healthy participants at average risk for colorectal cancer who have not undergone regular colon cancer screening.
* Determine participants' level of knowledge of this assessment.
* Determine participants' rate of acceptance into this study.

OUTLINE: This is a 2-part pilot study.

* Part 1: Participants complete a baseline questionnaire on attitudes, beliefs, and knowledge about colorectal cancer (CRC), CRC screening, and diet and genetic testing for colorectal cancer risk. Two-four weeks later, participants are educated about CRC screening options and undergo genetic and environmental risk assessment (GERA) decision counseling about the methylene tetrahydrofolate reductase (MTHFR) gene and dietary folate intake. Participants who decide to undergo GERA undergo blood testing for MTHFR polymorphisms and folate levels. Participants whose blood tests indicate low folate levels are further counseled about dietary folate intake.
* Part 2: Participants complete a questionnaire on attitudes, beliefs, and knowledge about CRC, CRC screening, and diet and genetic testing for colorectal cancer risk.

Participants in part 1 are followed at 1 week, 1 month, and then at 6 months.

PROJECTED ACCRUAL: A total of 110 participants (60 for part 1 and 50 for part 2) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Healthy participants
* Eligible for colorectal cancer screening
* No personal or family history of colorectal cancer

  * No more than 1 first-degree relative who has had colorectal cancer
* Part 1:

  * Has not undergone regular screening for colorectal cancer
* Part 2:

  * Not currently undergoing regular colon cancer testing, including any of the following:

    * Fecal occult blood testing within the past year
    * Flexible sigmoidoscopy or colonoscopy within the past 5 years

PATIENT CHARACTERISTICS:

Age

* 50 to 74

Performance status

* Not specified

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* Not specified

Renal

* Not specified

Other

* No inflammatory bowel disease (part 1 only)
* No concurrent health issues that would preclude study participation (part 1 only)
* No history of cancer except basal cell or squamous cell skin cancer (part 2 only)
* Able to speak and read English (part 2 only)

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* Not specified

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Not specified

Ages: 50 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Dates: Start 2003-11; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Colorectal cancer (CRC) screening rates by chart review at 4 months

SECONDARY OUTCOMES:
Knowledge regarding CRC risk by questionnaires at 4 and 12 months
CRC risk perception by questionnaires at 4 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: David Weinberg, MD, MSC, Study Chair — Fox Chase Cancer Center
Locations (4):
- United States (4):
  - Warren Grant Magnuson Clinical Center - NCI Clinical Studies Support, Bethesda, Maryland
  - Kimmel Cancer Center at Thomas Jefferson University - Philadelphia, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Vanderbilt-Ingram Cancer Center at Vanderbilt Medical Center, Nashville, Tennessee

REFERENCES:
- [Derived] Weinberg DS, Myers RE, Keenan E, Ruth K, Sifri R, Ziring B, Ross E, Manne SL. Genetic and environmental risk assessment and colorectal cancer screening in an average-risk population: a randomized trial. Ann Intern Med. 2014 Oct 21;161(8):537-45. doi: 10.7326/M14-0765. PMID 25329201